CLINICAL TRIAL: NCT06681103
Title: Online Personalized Normative Feedback to Foster Intention to Change and Help-Seeking in Young Adults With Gambling- and Trading-Related Problems: An Experimental Study
Brief Title: Online Intervention to Promote Change and Help-Seeking in Young Adults With Gambling and Trading Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Ministerio de Derechos Sociales, Consumo y Agenda 2030, Spain (Unknown)
Responsible Party: Principal Investigator, Ainhoa Coloma Carmona, PhD, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SUBV23/00004
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: This design follows a Solomon three-group structure, enabling the independent evaluation of the immediate effects that the pre-test assessment and the intervention may have on the study's dependent variables (intention to change and help-seeking behavior), as well as their maintenance three months after the intervention. The following experimental conditions will be established: (1) control group with pre- and post-test assessment (assessment group), (2) control group with post-test assessment only (delayed assessment group) and (3) intervention group with pre- and post-test assessment, which will also receive personalised online normative feedback on their gambling and trading behaviour after the initial assessment (PONF group). To adapt the PONF to each participant it is necessary to conduct a pre-test assessment, so an adaptation of Solomon's design will be used.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Online Normative Feedback (PONF) (Experimental): Participants in this group complete a pre-assessment measuring intention to change, help-seeking behavior, and gambling and trading behaviors (e.g., frequency and spending). They then receive personalized online normative feedback (PONF) based on their initial assessment and subsequently complete a post-assessment including the same outcomes.
  Within this intervention arm, participants are randomly assigned to one of two predefined assessment sequences (PNF-A vs. PNF-B), differing only in the timing of the post-intervention assessment of gambling and trading behaviors. This sequencing is implemented exclusively to support secondary analyses of potential reporting reactivity (e.g., social desirability) and does not involve any differences in intervention content, delivery, or assessment of the primary motivational outcomes.
  Interventions: Behavioral: Personalized Normative Feedback
- Control group 1 (Assessment group) (No Intervention): Participants in this group will complete both pre- and post-assessments on intention to change, help-seeking behavior, and gambling/trading behaviors. However, they will not receive any feedback. This group serves as a comparison to both intervention groups.
- Control group 2 (Delayed Assessment Group) (No Intervention): This group will complete only the post-assessment, measuring intention to change, help-seeking behavior, and gambling/trading behaviors, without completing a pre-test or receiving feedback, to independently analyze the immediate effects of the pre-test.

INTERVENTIONS:
Behavioral: Personalized Normative Feedback — Those participating in this condition will receive a personalised brief report which summarises the results of their initial assessment. The PONF will comprise the following elements: (1) Details of the main gambling and trading activities performed, including frequency of engagement and amount of money spent; (2) Scores on the criteria of pathological trading and/or PGSI (problem gambling), together with an interpretation of the results and the level of severity. All results will be accompanied by graphs enabling participants to compare their scores with the average scores of the Spanish population of the same sex and age range. To prevent an increase in behaviour in participants whose frequency or intensity of gambling/trading is below the norm, as recommended by Newall et al. (2023), the normative data will include extreme averages and percentages. All participants assigned to the PNF intervention receive identical feedback content, regardless of assessment sequencing.
  Arms: Personalized Online Normative Feedback (PONF)

SUMMARY:
The goal of this study is to investigate if personalized online normative feedback (PONF) can increase intention to change and help-seeking behaviors in young adults with gambling or trading problems in Spain. The main questions it aims to answer are:

1. Does PONF increase intention to change and help-seeking behaviors?
2. How does receiving PONF affect gambling and trading behaviors?

Researchers will compare three groups:

* Evaluation group: A control group with pre- and post-assessments.
* Delayed evaluation group: A control group with only a post-assessment, to control for the effect of the assessment.
* FNPO group: An intervention group receiving PONF after the initial evaluation and completing both pre- and post-assessments.

Participants will:

* Receive PONF or no feedback at the first evaluation.
* Complete initial and follow-up assessments after 12 weeks.

DETAILED DESCRIPTION:
Despite the availability of treatment options, the percentage of individuals with problem gambling who seek help or treatment remains low. To reach a larger number of pathological gamblers, other forms of online or self-guided interventions have been developed, with personalised normative feedback (NPF) being the most widely applied modality in the prevention of problem gambling in the young adult population. However, the majority of studies on the efficacy of PNF only assess its impact on the intensity and severity of gambling behaviour, and do not analyse its potential effect on increasing intention to change and treatment-seeking behaviour. Furthermore, there is a lack of studies analyzing the efficacy of NPF in reducing new forms of online money spending linked to pathological gambling, such as betting on video games and excessive trading of financial assets, including cryptocurrencies.

The present project has two objectives: (1) to quantify the intention to change and the prevalence of help-seeking behaviours in the Spanish young adult population with pathological gambling or trading behaviours; and (2) to analyze the effectiveness of personalised online normative feedback (PONF) to increase intention to change and help-seeking in this population.

The study will employ a randomised controlled design (three Solomon groups) with one intervention group and two control groups. The study will involve a sample of at least 656 men and women living in Spain, aged between 18 and 34 years. The impact of receiving FNPO on gambling and trading behaviour will be analysed over a 12-week period. This will include an assessment of the intention to change and treatment seeking, as well as the longitudinal trajectory of gambling and trading behaviours (in terms of intensity, frequency and severity). Furthermore, individual, interpersonal and contextual factors will be evaluated in order to ascertain the profile of those with gambling and trading issues who may derive the greatest benefit from this type of intervention.

This project is pioneering both nationally and internationally. Furthermore, this study will assess for the first time the intention to change and help-seeking in young adults with gambling behaviour (in traditional and new formats such as video games) and pathological trading. It will also develop and analyze the effectiveness of the first tool to mobilize change and reduce the prevalence of these behaviours. Furthermore, the study design will enable an independent assessment of the impact of both the intervention and the assessment of pathological gambling and trading behaviours on the individual.

ELIGIBILITY:
Participants' eligibility will be assessed based on sociodemographic variables and measures of psychological distress, suicidal behavior, sleep quality and substance use. Eligible participants for the study on PONF's effect on intention to change and help-seeking behavior in young adults with gambling or trading problems must meet the following inclusion and exclusion criteria.

Inclusion Criteria:

* Engaged in trading or gambling activities (land-based or online) at least once per month in the past 60 days
* Aged 18-34 years
* Residing in Spain
* Provide informed consent to participate in initial online assessment, post-test, and follow-up

Exclusion Criteria:

* Currently undergoing psychological or psychiatric treatment
* Scoring above 3 on the Oviedo Infrequency Scale (Fonseca-Pedrero et al., 2009), indicating potential random/pseudorandom or dishonest responses.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1112 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Intention to change | Baseline, immediate follow-up (after PONF), 3-month follow-up
  The study will assess intention to change and help-seeking behavior using three custom items. In the initial assessment, participants will respond to a dichotomous question regarding whether they have considered reducing or abandoning gambling/trading in the past year. They will also rate the likelihood of engaging in these behaviors over the next 12 months on a scale from 0% (not likely) to 100% (very likely). Finally, participants will indicate their goal regarding their gambling/trading behavior, choosing from options to reduce, increase, maintain, or cease the behavior.
Treatment-seeking behavior | Baseline, immediate follow-up (after PONF), 3-month follow-up
  Treatment-seeking behavior will be assessed during the initial evaluation using a the following question: "Have you ever sought professional help, advice from family or friends, or done something on your own to limit or reduce your [gambling/trading] behavior?" If participants answer "yes," they will complete the Help-Seeking Questionnaire (HSQ), which includes 14 items assessing in-person (e.g., seeing a psychologist), remote (e.g., calling a helpline), and self-directed (e.g., reading forums or searching websites) help-seeking behaviors.

SECONDARY OUTCOMES:
Gambling and trading behaviors | Baseline, immediate follow-up (after PONF), 3-month follow-up
  The frequency and intensity of gambling and trading behaviors will be assessed with ad-hoc items. Gambling behavior will be evaluated with reference to the last year during the initial and post-test assessments, and for the last month during the 3-month follow-up. Trading behavior will focus on financial operations, types of trading, and frequency of market monitoring. A dichotomous item will also assess whether participants engage in professional or amateur trading.
Disordered gambling | Baseline, 3-month follow-up
  The Problem Gambling Severity Index (PGSI) and the Gambling Disorder Identification Test (GDIT) will be used to assess problem gambling. The Problem Gambling Severity Index (9 items) categorises participants as non-problem, low-risk, moderate-risk, or problem gambling. The total score ranges from 0 to 27, with higher scores indicating a greater severity of gambling problems.
  The investigators will adapt the Gambling Disorder Identification Test, a 14-item Likert scale, to Spanish and validate it as a new measure. It evaluates gambling behaviours, symptoms, and negative consequences, categorising participants as non-gamblers, recreational gamblers, or problematic gamblers (mild, moderate, severe). The total score of the scale ranges from 0 to 62, with higher scores indicating more severe gambling disorder.
Disordered trading | Baseline, 3-month follow-up
  Trading Disorder Scale which is based on the diagnostic criteria for gambling disorder from the DSM-5, adapted to evaluate problematic trading behaviors. This scale evaluates various dimensions of addictive behavior, including tolerance, withdrawal, loss of control, craving, social impairment, and continued engagement despite negative consequences. The total score of the scale ranges from 0 to 13, with scores ≥5 indicates the possible presence of disordered trading.

OTHER OUTCOMES:
Gambling and trading-related harms | Baseline and 3-month follow-up
  An adapted version of the Short Gambling Harm Screen will be used to evaluate harms related to both gambling and trading activities, employing a yes/no response format. Scores range from 0 to 10, with higher scores indicating greater gambling/trading-related harm.
Gambling and trading self-efficacy | Baseline and 3-month follow-up
  The Brief Situational Questionnaire, adapted for gambling and trading behaviors, will assess self-efficacy in resisting gambling or trading across 10 specific scenarios. Scores range from 0 to 100, reflecting the degree of self-efficacy to resist these behaviors, with higher scores indicating stronger self-efficacy in handling such situations.
Peer gambling and trading | Baseline
  It will be assessed using a custom dichotomous item (yes/no) that evaluates whether the participant's friends or family engage in gambling, trading or financial investments.
Satisfaction and perceived usefulness | Immediate follow-up
  Feedback on the satisfaction with the personalized normative feedback received and the perceived usefulness of the information provided will be assessed using a 4-point Likert questionnaire (only in intervention groups). Scores range from 1 to 4, with higher scores reflect greater satisfaction and perceived usefulness of the PONF.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Hernández University, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No